CLINICAL TRIAL: NCT00674531
Title: Detection of Enterovirus RNA by RT-PCR in Atheromatous Lesions
Brief Title: Detection of Enterovirus RNA in Atheromatous Lesions
Acronym: ATH-ENTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0608071; 2007-A00895-48 (Other: AFSSAPS); DGS2007-0534 (Other: DGS)
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Arteriosclerosis
Keywords: Arteriosclerosis; Arterial Occlusive Diseases; Enterovirus; Artery resection
MeSH Terms: conditions — Arteriosclerosis; Arterial Occlusive Diseases; Enterovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Enterovirus RNA analysis
  Interventions: Procedure: Artery resection

INTERVENTIONS:
Procedure: Artery resection — Artery resection

SUMMARY:
Atherosclerosis is one of the first causes of morbidity-mortality in industrialized countries. Numerous works suggest that some infectious agents could be involved in the inflammatory process leading to the development of this pathology, such as Chlamydophila pneumoniae, cytomegalovirus or herpes simplex virus. Enteroviruses are small RNA viruses that have been incriminated in various acute or chronic cardiac diseases (pericarditis, myocarditis, dilated cardiomyopathy) and exhibit a tropism for vascular endothelia. Different clinical and experimental arguments suggest that they could play a cofactor role in the occurrence or maintenance of atherosclerosis lesions. A multicenter study developed in collaboration with colleagues of the University Hospital of Reims (France) showed that it was frequent to detect enterovirus RNA in cardiac biopsies from patients with myocardial infarction. Furthermore, a pilot study conducted in the University Hospital of Saint-Etienne (France) on atheromatous arterial samples from 18 patients allowed the detection of enterovirus RNA in 20% of them.

DETAILED DESCRIPTION:
Objective: In order to complete these data and to answer clearly to the question of the role of persistent infection by enteroviruses in atherosclerosis, we propose this research program involving the Departments of Vascular Surgery of three University hospitals of the "Rhône-Alpes" region and of three laboratories of Virology interested by the relationship between chronic diseases and enterovirus infection..

Methods: It is projected to include about one hundred voluntary adults exhibiting carotid atheromatous lesions requiring a surgical removal. Because of the difficulty to define a pertinent control group, each patient will be his/her own control. In addition to the fragment of pathologic carotid, it will be taken arterial and venous fragments from vessels that are never the seat of atherosclerosis lesions. To reach the best sensitivity, enterovirus RNA will be detected by nested RT-PCR.

Evaluation criteria: The main evaluation criterion will be the percentage of detection of enterovirus RNA by RT-PCR in atheromatous lesions by comparison to control arteries by Mac-Nemar test. These results will be correlated to anatomic and histological lesions of the atheromatous plaques. Other markers will be analysed secondarily: detection of enterovirus RNA in control venous samples, detection of stigmata of viral replication by immunochemistry or detection of negative RNA strands, analysis of the antibody response to enterovirus in blood, molecular typing of enteroviruses detected in the lesions… Expected benefits: This study should allow to better understand the putative involvement of enteroviruses in atherosclerosis-linked diseases. If the hypothesis of a relationship was confirmed, a more ambitious research project would be proposed in order to investigate the mechanisms by which enterovirus can favour atherosclerosis and to discuss the opportunity of preventive strategies (notably vaccination) to reduce the risk.

ELIGIBILITY:
Inclusion Criteria:

* Indication of artery resection
* affiliated or a beneficiary of a social security category
* having signed the inform consent form

Exclusion Criteria:

* pregnant women
* contra-indication to clamping
* scheduled resection at friday after-noon, week-end or legal holidays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Prévalence of detection of enteroviral RNA by RT-PCR in atherosclerotic carotid artery in comparison with sound carotid artery | artery resection

SECONDARY OUTCOMES:
Prevalence of detection of enteroviral RNA by RT-PCR in atherosclerotic carotid artery in comparison with sound vein | Artery resection
Prevalence of detection of enteroviral RNA by RT-PCR in sound carotid artery in comparison with sound vein | Artery resection
Prevalence of detection of enteroviral RNA by RT-PCR in calm and active atherosclerotic lesions | Artery resection
Prevalence of detection of antibodies between different groups of patients. | Artery resection
Prevalence of detection of enteroviral RNA by RT-PCR in atherosclerotic carotid artery in comparison with circulating blood | Artery resection

CONTACTS AND LOCATIONS:
Overall Officials: Xavier BARRAL, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CHU de Saint-Etienne, Saint-Etienne

REFERENCES:
- [Background] Schanen C, Nasri D, Bourlet T, Barral X, Favre JP, Bourrat D, Peoc'h M, Ginevra C, Andreoletti L, Pozzetto B, Pillet S. Enterovirus in arteriosclerosis: a pilot study. J Clin Virol. 2007 Jun;39(2):106-12. doi: 10.1016/j.jcv.2007.03.014. Epub 2007 May 10. PMID 17499019
- [Background] Andreoletti L, Venteo L, Douche-Aourik F, Canas F, Lorin de la Grandmaison G, Jacques J, Moret H, Jovenin N, Mosnier JF, Matta M, Duband S, Pluot M, Pozzetto B, Bourlet T. Active Coxsackieviral B infection is associated with disruption of dystrophin in endomyocardial tissue of patients who died suddenly of acute myocardial infarction. J Am Coll Cardiol. 2007 Dec 4;50(23):2207-14. doi: 10.1016/j.jacc.2007.07.080. Epub 2007 Nov 19. PMID 18061067